CLINICAL TRIAL: NCT01957163
Title: A Study to Compare the Addition of Umeclidinium Bromide (UMEC) to Fluticasone Furoate (FF)/Vilanterol (VI), With Placebo Plus FF/VI in Subjects With Chronic Obstructive Pulmonary Disease (COPD) -Study 1
Brief Title: Study to Compare the Addition of Umeclidinium Bromide (UMEC) to Fluticasone Furoate (FF)/Vilanterol (VI), With Placebo Plus FF/VI in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200109
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Results first posted 2014-11-25 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: dry powder inhaler; fluticasone furoate/vilanterol; umeclidinium bromide; safety; long acting beta2- receptor agonist; long acting muscarininc receptor antagonist; efficacy; COPD; inhaled corticosteroid
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- FF/VI 100/25 mcg + UMEC (62.5mcg) (Experimental): Subjects received one inhalation of FF/VI 100/25 mcg via a DPI followed by one inhalation UMEC (62.5mcg) via DPI once-daily in the morning for 12 weeks.
  Interventions: Drug: FF; Drug: VI; Drug: UMEC
- FF/VI 100/25 mcg + UMEC (125mcg) (Experimental): Subjects received one inhalation of FF/VI 100/25 mcg via DPI followed by one inhalation of UMEC (125mcg) via a DPI once-daily in the morning for 12 weeks.
  Interventions: Drug: FF; Drug: VI; Drug: UMEC
- FF/VI 100/25 mcg + Placebo (Experimental): Subjects received one inhalation of FF/VI 100/25 mcg via DPI followed by one inhalation of matching placebo via a DPI once-daily in the morning for 12 weeks.
  Interventions: Drug: FF; Drug: VI; Drug: Placebo

INTERVENTIONS:
Drug: FF — Dry white powder containing 100mcg of Fluticasone Furoate blended with lactose per blister was administered by DPI.
Drug: VI — Dry white powder containing 25mcg of Vilanterol micronised drug (as the 'M' salt triphenylacetate) blended with lactose and magnesium stearate per blister was administered by DPI.
Drug: UMEC — Umeclidinium bromide in a powder blend with lactose and magnesium stearate was used at two different doses 62.5mcg and 125mcg.
  Arms: FF/VI 100/25 mcg + UMEC (125mcg); FF/VI 100/25 mcg + UMEC (62.5mcg)
Drug: Placebo — The matching placebo DPI identical in appearance to the inhaler containing active study medication.
  Arms: FF/VI 100/25 mcg + Placebo

SUMMARY:
After screening, subjects will enter a 4 week open-label run-in period with fluticasone furoate (FF)/vilanterol (VI) 100/25 mcg administered once daily via dry powder inhaler (DPI). Subjects will then be randomized to receive any one of the 3 treatments (umeclidinium bromide [UMEC] [62.5 mcg] administered once daily via a DPI; OR UMEC [125 mcg] administered once daily via a DPI; OR matching placebo administered once daily via a DPI), while continuing treatment with open label FF/VI 100/25 mcg during a 12-week treatment period. There will be a total of eight scheduled clinic visits at Pre-Screening (Visit0), Screening (Visit 1), blinded treatment Day 1(Visit2), 2(Visit3), 28 (Visit4), 56 (Visit5), 84 (Visit6) and 85 (Visit7). A follow-up phone contact will be conducted approximately 7 days after the last clinic visit. The total duration of subject participation in the study from Screening to Follow-up will be approximately 17 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed Consent: A signed and dated written informed consent prior to study participation.
* Age: Subjects 40 years of age or older at Visit 1.
* Gender: Male or female subjects.
* A female is eligible to enter and participate in the study if she is of:
* Non-child bearing potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile). Surgically sterile females are defined as those with a documented hysterectomy and/or bilateral oophorectomy or tubal ligation. Post-menopausal females are defined as being amenorrhoeic for greater than 1 year with an appropriate clinical profile, e.g., age appropriate, >45 years, in the absence of hormone replacement therapy.

OR

* Child bearing potential, has a negative pregnancy test at screening, and agrees to one of the following acceptable contraceptive methods used consistently and correctly (i.e., in accordance with the approved product label and the instructions of the physician for the duration of the study - screening to follow-up contact):
* Abstinence
* Oral Contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) that meets the SOP effectiveness criteria as stated in the product label
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject. For this definition, "documented" refers to the outcome of the investigator's/designee's medical examination of the subject or review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records.
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)
* Diagnosis: An established clinical history of COPD in accordance with the definition by the American Thoracic Society/European Respiratory Society.
* Smoking History: Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years [number of pack years = (number of cigarettes per day / 20) x number of years smoked (e.g., 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack year history.
* Severity of Disease: A pre and post-albuterol/salbutamol FEV1/FVC ratio of <0.70 and a pre and post-albuterol/salbutamol FEV1 of <=70% of predicted normal values at Visit 1 (Screening) calculated using Nutrition Health and Examination Survey (NHANES) III reference equations.
* Dyspnea: A score of >=2 on the mMRC Dyspnea Scale at Visit 1.
* QTc Criteria:
* QTc(F) <450 milliseconds (msec) or
* QTc(F) <480msec for patients with QRS duration >=120msec
* The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB), Fridericia's formula (QTcF), or another method, machine or manual overread.
* For subject eligibility and withdrawal, QTcF will be used.
* For purposes of data analysis, QTcF will be used as primary.
* The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating or are planning on becoming pregnant during the study.
* Asthma: A current diagnosis of asthma.
* Other Respiratory Disorders: Known alpha-1 antitrypsin deficiency, active lung infections (such as tuberculosis), and lung cancer are absolute exclusionary conditions. A subject who, in the opinion of the investigator, has any other significant respiratory conditions in addition to COPD should be excluded. Examples may include clinically significant bronchiectasis, pulmonary hypertension, sarcoidosis, or interstitial lung disease.
* Other Diseases/Abnormalities: Subjects with historical or current evidence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or hematological abnormalities that are uncontrolled and/or a previous history of cancer in remission for <5 years prior to Visit 1 (localized carcinoma of the skin that has been resected for cure is not exclusionary). Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the efficacy or safety analysis if the disease/condition exacerbated during the study.
* Contraindications: Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, beta2-agonist, sympathomimetic, corticosteroid (intranasal, inhaled or systemic) lactose/milk protein or magnesium stearate, or a medical condition such as narrow-angle glaucoma, prostatic hypertrophy or bladder neck obstruction, that, in the opinion of the study physician contraindicates study participation or use of an inhaled Long acting muscarinic antagonist (LAMA), Long acting beta agonist (LABA) or Inhaled corticosteroids (ICS).
* Hospitalization: Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1.
* Lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to Visit 1.
* Lung Resection: Subjects with lung volume reduction surgery within the 12 months prior to Visit 1.
* 12-Lead ECG: An abnormal and clinical significant ECG finding from the 12-lead ECG conducted at Visit 1. Investigators will be provided with ECG reviews conducted by a centralized independent cardiologist to assist in evaluation of subject eligibility. The study investigator will determine the medical significance of any ECG abnormalities.
* Clinically significant and abnormal laboratory finding at Screening (Visit1). After discussion with the Medical Monitor, the investigator may have the option to verify the abnormal lab result prior to Visit2
* Medication Prior to Spirometry: Unable to withhold albuterol/salbutamol for the 4 hour period required prior to spirometry testing at each study visit.
* Excluded Medications: Use of the following medications are not permitted within the defined time intervals prior to Visit 1and throughout the study:
* No use within 12 weeks prior to Screening Visit 1 or thereafter at any time during the study: Depot corticosteroids.
* No use within 6 weeks prior to Screening Visit 1 or thereafter at any time during the study: Systemic, oral or parenteral corticosteroids (Intra-articular corticosteroid injections are permitted.), Antibiotics (for lower respiratory tract infection), Cytochrome P450 3A4 strong inhibitors.
* No use within 14 days prior to Screening Visit 1 or thereafter at any time during the study: Phosphodiesterase 4 inhibitors (roflumilast).
* No use within 10 days prior to Screening Visit 1 or thereafter at any time during the study: Olodaterol and Indacaterol.
* No use within 7 days prior to Screening Visit 1 or thereafter at any time during the study: Long acting muscarinici antagonists (tiotropium, aclidinium, glycopyrronium).
* No use within 48 hrs prior to Screening Visit 1 or thereafter at any time during the study: Theophyllines, Oral leukotriene inhibitors (zafirlukast, montelukast, zileuton), Salmeterol and formoterol, ICS/LABA combinations (e.g., fluticasone propionate/salmeterol, mometasone furoate/formoterol fumarate, budesonide/formoterol fumarate), Oral beta2-agonists Long-acting.
* No use within 24 hrs prior to Screening Visit 1 or thereafter at any time during the study: Inhaled sodium cromoglycate or nedocromil sodium.
* No use within 12 hrs prior to Screening Visit 1 or thereafter at any time during the study: Oral beta2-agonists Short-acting.
* No use within 4 hrs prior to Screening Visit 1 or thereafter at any time during the study: Inhaled short acting beta2-agonists (use of study provided prn albuterol/salbutamol is permitted during the study, except in the 4-hour period prior to spirometry testing.), Inhaled short-acting anticholinergics, Inhaled short-acting anticholinergic/short-acting beta2-agonist combination products.
* No use within 30 days or 5 half lives whichever is longer prior to Screening Visit 1 or thereafter at any time during the study: Any other investigational drug.
* Prior enrolment in one of the replicate studies: subjects who have previously been assigned a subject number (enrolled) in study 200110 that is a replicate study of 200109.
* Oxygen: Use of long-term oxygen therapy (LTOT) described as oxygen therapy prescribed for greater than 12 hours a day. As-needed oxygen use (i.e., <=12 hours per day) is not exclusionary.
* Nebulized Therapy: Regular use (prescribed for use every day, not for as-needed use) of short-acting bronchodilators (e.g., albuterol/salbutamol) via nebulized therapy.
* Pulmonary Rehabilitation Program: Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Visit 1, or who will enter the acute phase of a pulmonary rehabilitation program during the study. Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded.
* Drug or Alcohol Abuse: A known or suspected history of alcohol or drug abuse within 2 years prior to Visit 1.
* Affiliation with Investigator Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Inability to read: In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 619 (Actual)
Dates: Start 2013-10-01; Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- United States (13):
  - GSK Investigational Site, Jasper, Alabama
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Morgantown, West Virginia
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Canada (10):
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Greater Sudbury, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Gatineau, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, St-Romulad, Quebec
- Chile (7):
  - GSK Investigational Site, Quillota, Región de Valparaíso
  - GSK Investigational Site, Concepción, Región Del Biobio
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talca, Región Metro de Santiago
  - GSK Investigational Site, Santiago
  - GSK Investigational Site, Viña del Mar
- Romania (7):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Codlea
  - GSK Investigational Site, Râmnicu Vâlcea
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 200109 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200109 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200109 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200109 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200109 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200109 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200109 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants ≥ 40 years of age with history of chronic obstructive pulmonary disease (COPD) and a smoking history of ≥ 10 pack-years were enrolled in the study. Participants completed a 4-week run-in period, in which they received fluticasone furoate 100 micrograms(µg)/vilanterol 25 µg, followed by a 12-week treatment period and 1-week follow-up.
Pre-assignment Details: A total of 619 participants (pars.), representing the enrolled particpants, were randomized to study treatment and comprised the Intent-to-Treat (ITT) Population (participants randomized to treatment who received ≥ 1 dose of randomized study medication in the treatment period).
Groups:
- FF/VI 100/25 µg + Placebo: Participants received one inhalation of fluticasone furoate/vilanterol (FF/VI) 100/25 µg once-daily (OD) via a dry powder inhaler (DPI), followed by one inhalation of umeclidinium bromide (UMEC) matching placebo, administered via a dry powder inahler in the morning for 12weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study, for symptomatic relief from COPD symptoms.
- FF/VI 100/25 µg + UMEC 62.5 µg: Participants received one inhalation of fluticasone furoate/vilanterol 100/25 µg once- daily via a dry powder inhalerfollowed by one inhalation of umeclidinium bromide 62.5 µg administered via a dry powder inhaler in the morning for 12weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study, for symptomatic relief from COPD symptoms.
- FF/VI 100/25 µg + UMEC 125 µg: Participants received one inhalation of fluticasone furoate/vilanterol 100/25 µg once- daily via a dry powder inhaler followed by one inhalation of umeclidinium bromide 125 µg administered via a dry powder inhaler in the morning for 12 weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study, for symptomatic relief from COPD symptoms.
Period: Overall Study
Arm/Group | FF/VI 100/25 µg + Placebo | FF/VI 100/25 µg + UMEC 62.5 µg | FF/VI 100/25 µg + UMEC 125 µg
Started | 206 | 206 | 207
Completed | 191 | 195 | 189
Not Completed | 15 | 11 | 18
Not completed — Adverse Event | 5 | 2 | 4
Not completed — Lack of Efficacy | 5 | 4 | 9
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Met Protocol-Defined Stopping Criteria | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- FF/VI 100/25 µg + Placebo: Participants received one inhalation of fluticasone furoate/vilanterol 100/25 µg OD via a DPI, followed by one inhalation of UMEC matching placebo, administered via a DPI in the morning for 12weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study, for symptomatic relief from COPD symptoms.
- FF/VI 100/25 µg + UMEC 62.5 µg: Participants received one inhalation of fluticasone furoate/vilanterol 100/25 µg OD via a DPI followed by one inhalation of UMEC 62.5 µg administered via a DPI in the morning for 12weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study, for symptomatic relief from COPD symptoms.
- FF/VI 100/25 µg + UMEC 125 µg: Participants received one inhalation of fluticasone furoate/vilanterol 100/25 µg OD via a DPI followed by one inhalation of UMEC 125 µg administered via a DPI in the morning for 12 weeks. In addition, participants were provided supplemental albuterol/salbutamol inhalation aerosol to be used as needed throughout the study, for symptomatic relief from COPD symptoms.
- Total: Total of all reporting groups
Arm/Group | FF/VI 100/25 µg + Placebo | FF/VI 100/25 µg + UMEC 62.5 µg | FF/VI 100/25 µg + UMEC 125 µg | Total
Number analyzed (Participants) | 206 | 206 | 207 | 619
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (7.90) | 64.9 (8.72) | 63.8 (7.65) | 64.4 (8.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 80 | 212
  Male | 141 | 139 | 127 | 407
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 5 | 4 | 5 | 14
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  White - Arabic/North African Heritage | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 200 | 201 | 202 | 603

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Trough Forced Expiratory Volume in One Second (FEV1) at Day 85
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 on Day 85 is defined as the mean of the FEV1 values obtained 23 and 24 hours after dosing on Day 84. Analysis was performed using a mixed model repeated measures (MMRM) with covariates of treatment, Baseline FEV1, smoking status, Day, treatment, Day by baseline interaction and Day by treatment interaction, Day being nominal. Baseline FEV1 is the mean of the two assessments made at 30 and 5 minutes (min) pre-dose on Day 1. The change from baseline value is the difference between the on-treatment value and the baseline value.
Time Frame: Day 85
Population: ITT Population: all pars. randomized to treatment who received ≥ 1 dose of randomized study medication in the Treatment Period. Number of pars. presented represent those with data available at given time point; however, all pars. in the ITT population without missing covariate information, with ≥ 1 post BL measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 µg + Placebo | FF/VI 100/25 µg + UMEC 62.5 µg | FF/VI 100/25 µg + UMEC 125 µg
Number analyzed (Participants) | 190 | 195 | 188
Liters | -0.020 (0.0111) | 0.103 (0.0110) | 0.108 (0.0111)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg + Placebo vs FF/VI 100/25 µg + UMEC 62.5 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measure; Restricted maximum likelihood (REM) - based repeated measure approach (MMRM); Least squared mean difference = 0.124, 95% CI 2-sided [0.093 to 0.154]
Statistical Analysis 2: Comparison: FF/VI 100/25 µg + Placebo vs FF/VI 100/25 µg + UMEC 125 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measure; Restricted maximum likelihood (REM) - based repeated measure approach (MMRM); Least squared mean difference = 0.128, 95% CI 2-sided [0.098 to 0.159]

2. Secondary Outcome: Change From Baseline in Weighted Mean (WM), 0-6 Hour FEV1 Obtained Post-dose at Day 84
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. The 0-6 hour weighted mean was derived by calculating the area under the FEV1/time curve over the nominal time points of 0 hour (trough value), 15 and 30 min, 1, 3 and 6 hours, using the trapezoidal rule, and then dividing by the actual time between dosing and the 6 hour assessment. Analysis was performed using MMRM with covariates of treatment, Baseline FEV1 (mean of the two assessments made 30 minutes and 5 minutes pre-dose on Day 1), smoking status, Day, and Day by Baseline and Day by treatment interactions. Baseline FEV1 is the mean of the two assessments made at 30 and 5 min pre-dose on Day 1. The change from baseline value is the difference between the on-treatment value and the baseline value.
Time Frame: Day 84
Population: ITT Population. Number of participants presented represent those with data available at the time point being presented; however, all participants in the ITT population without missing covariate information and with at least one post baseline measurement are included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF/VI 100/25 µg + Placebo | FF/VI 100/25 µg + UMEC 62.5 µg | FF/VI 100/25 µg + UMEC 125 µg
Number analyzed (Participants) | 191 | 195 | 189
Liters | 0.034 (0.0123) | 0.187 (0.0122) | 0.175 (0.0123)
Statistical Analysis 1: Comparison: FF/VI 100/25 µg + Placebo vs FF/VI 100/25 µg + UMEC 125 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measure; Restricted maximum likelihood (REM) - based repeated measure approach (MMRM); Least squared mean difference = 0.153, 95% CI 2-sided [0.118 to 0.187]
Statistical Analysis 2: Comparison: FF/VI 100/25 µg + Placebo vs FF/VI 100/25 µg + UMEC 125 µg; Test type: Superiority or Other; p < 0.001, Mixed Model Repeated Measure; Restricted maximum likelihood (REM) - based repeated measure approach (MMRM); Least squared mean difference = 0.140, 95% CI 2-sided [0.106 to 0.175]

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from start of study medication until follow-up visit (up to 14 weeks)
Description: On-treatment SAEs and non-serious AEs are reported for members of the ITT Population, comprised of all participants randomized to treatment who received at least one dose of randomized study medication in the treatment period.
Arm/Group | FF/VI 100/25 µg + Placebo | FF/VI 100/25 µg + UMEC 62.5 µg | FF/VI 100/25 µg + UMEC 125 µg
Serious Adverse Events (participants affected / at risk) | 6/206 | 2/206 | 7/207
Other Adverse Events (participants affected / at risk) | 15/206 | 26/206 | 26/207
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg + Placebo (N=206) | FF/VI 100/25 µg + UMEC 62.5 µg (N=206) | FF/VI 100/25 µg + UMEC 125 µg (N=207)
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4
Pneumonia (Infections and infestations) | 2 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 0 | 1
Shunt stenosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF/VI 100/25 µg + Placebo (N=206) | FF/VI 100/25 µg + UMEC 62.5 µg (N=206) | FF/VI 100/25 µg + UMEC 125 µg (N=207)
Nasopharyngitis (Infections and infestations) | 7 | 7 | 10
Headache (Nervous system disorders) | 6 | 9 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 7 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.